CLINICAL TRIAL: NCT03284697
Title: Success of Direct Pulp Capping With Mineral Trioxide Aggregate and Calcium Hydroxide In Cariously Exposed Teeth: A Randomized Clinical Study.
Brief Title: Direct Pulp Capping With MTA and Calcium Hydroxide.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Principal, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Komal Suhag
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Reversible Pulpitis
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPC with Ca(OH)2 (Active Comparator): Direct pulp capping with Ca(OH)2.
  Interventions: Procedure: Direct Pulp Capping with Ca(OH)2
- DPC with MTA (Active Comparator): Direct pulp capping with MTA
  Interventions: Procedure: Direct Pulp Capping With MTA

INTERVENTIONS:
Procedure: Direct Pulp Capping with Ca(OH)2 — Calcium hydroxide powder was mixed with saline and placed over the exposed pulp tissue. The cavities were then restored with resin modified GIC liner followed by composite restoration.
  Other Names: Vital Pulp Therapy
  Arms: DPC with Ca(OH)2
Procedure: Direct Pulp Capping With MTA — MTA was mixed using1:3 water/ powder ratio and applied to exposure site. Then cotton pellets soaked in normal saline was placed over MTA and cavity was sealed provisionally with IRM. After 24 hours, the patient was recalled and the cavity was restored with resin modified GIC liner followed by composite restoration.
  Other Names: Vital pulp therapy
  Arms: DPC with MTA

SUMMARY:
Aim of the study was to evaluate and compare clinical and radiographic success with MTA and calcium hydroxide as direct pulp capping materials in cariously exposed mandibular molars.

Study was conducted in Post Graduate Institute of Dental Sciences, Rohtak in department of Conservative Dentistry & Endodontics. Mature permanent mandibular molars with reversible pulpitis exhibiting occlusal pulp exposure from primary dental caries were included in the study. After excavation of caries and obtaining pulpal hemostasis, patients were randomly allocated into two groups- MTA and Calcium Hydroxide. Pulp was capped with respective allocated material and then tooth in both groups were restored according to standard protocol.

DETAILED DESCRIPTION:
AIM AND OBJECTIVES The present study aims to

1. Evaluate the success of direct pulp capping in mandibular molar teeth.
2. Evaluate and compare the clinical and radiographic success with MTA and calcium hydroxide as direct pulp capping materials.
3. To assess the pain intensity before and after the direct pulp capping with visual analog scale (VAS).

MATERIALS AND METHODS Study subjects were recruited from the patients visiting the Department of conservative dentistry and endodontics, PGIDS, Rohtak.

METHODOLOGY Prior to treatment, a thorough clinical and radiological examination was carried out.

A thorough history will be taken from each patient. Prior informed consent was obtained either from the patient or guardians after explaining the procedure, risks and benefits.

Clinical procedure:

Mature mandibular permanent molars exhibiting deep caries approaching pulp were chosen for the study.

The teeth were evaluated by periapical radiographs, periodontal probing, percussion test, and vitality assessment with thermal test and electric pulp test; the teeth determined to have reversible pulpitis were included.

All periapical radiographs were exposed by using constant kVP, mA, and exposure time (70 KVP, 8 mA, and 0.8 sec.) with a Rinn paralleling device and processed manually.

After administration of local anesthesia, rubber dam isolation of the involved tooth was done.

The tooth was disinfected by scrubbing with 2% chlorhexidine and 75% isopropyl alcohol.

Initially caries was removed with round bur under sterile water spray. Then, the remaining caries was removed carefully with a spoon excavator. After complete caries excavation, disinfection of exposed pulp with 2.5% sodium hypochlorite irrigation and a soaked cotton pellet was done.

Then sodium hypochlorite dressing was placed for 10 minutes to achieve adequate pulpal hemostasis.

Patients were randomly allocated into two groups (Group I - MTA and Group II -Calcium hydroxide) using a computer program This study was a double blinded trial i.e. both the patient and the investigator were not aware of the group to which the participant belongs.

GROUP I- CALCIUM HYDROXIDE GROUP Calcium hydroxide powder was mixed according to manufacturer's instructions and applied directly onto the exposed pulps.

The cavities were then restored with resin modified GIC liner followed by composite restoration.

GROUP II - MTA GROUP MTA was mixed according to manufacturer's instructions i.e. 1:3 water/ powder ratio and applied to exposure site with a sterile carrier.

Then cotton pellets soaked in normal saline was placed over MTA and cavity was sealed temporarily with intermediate restoration material.

After 24 hours, the patient was recalled and the setting of MTA was confirmed and the cavity was restored with resin modified GIC liner followed by composite restoration.

FOLLOW UP The patients were recalled periodically at 1 week, 3 months, 6 months and 12 months after the direct pulp capping procedure for clinical (post operative sensitivity, pain, tenderness, vitality) and radiographic (widening of periodontal ligament space and periapical radiolucency) evaluation.

CRITERIA FOR SUCCESSFUL OUTCOME A positive vitality test. No pain on percussion. No widening of periodontal ligament on periapical radiograph. No clinical or radiographic signs and/or symptoms of irreversible pulpitis and pulp necrosis.

CRITERIA FOR FAILURE No response to pulp vitality test. Teeth exhibiting clinical or radiographic signs and/or symptoms of irreversible pulpitis and pulp necrosis.

Postoperative pain assessment:

This was done using Horizontal VAS scale preoperatively, 6, 12, 18 hours, 1, 2, 3, 4, 5, 6, and 7 days after the procedure.

The pain VAS was completed by the patients themselves. The patients were asked to place a line perpendicular to the VAS line at the point that represents their pain intensity.

Patients were also asked to take analgesic (ibuprofen 400 mg/6-8h) according to the intensity of pain experienced by them and note down the details of analgesic intake on the proforma regarding the number of doses required and timing of the dose.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to participate in the study.
* Age group- 15-40 years.
* Mature permanent mandibular molars with reversible pulpitis.
* Teeth exhibiting occlusal pulp exposure from primary dental caries.

Exclusion Criteria:

* Primary teeth.
* Teeth with irreversible pulpitis (spontaneous pain) or pulp necrosis, chronic periodontitis, cracked tooth, internal or external resorption, calcified canals, associated with sinus tract, and furcation or apical radiolucency.
* Immuno-compromised, diabetic, pregnant and hypertensive patients.
* Positive history of antibiotic and analgesic use within past one month of the treatment.
* Failure to obtain authorization from patients.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate and compare the clinical and radiographic success with MTA and calcium hydroxide as direct pulp capping materials. | Baseline to 1 year
  CRITERIA FOR SUCCESSFUL OUTCOME
  * A positive vitality test.
  * No pain on percussion.
  * No widening of periodontal ligament on periapical radiograph.
  * No clinical or radiographic signs and/or symptoms of irreversible pulpitis and pulp necrosis.
  CRITERIA FOR FAILURE
  * No response to pulp vitality test.
  * Teeth exhibiting clinical or radiographic signs and/or symptoms of irreversible pulpitis and pulp necrosis.

SECONDARY OUTCOMES:
To assess the pain intensity before and after the direct pulp capping with visual analog scale (VAS). | Baseline to 7 days
  Patients were instructed to score the pain experienced by them using VAS scale. Pain was recorded preoperatively, 6, 12, 18 hours, 1, 2, 3, 4, 5, 6, and 7 days following the procedure.
  Pain intensity was categorized as: no pain (0 - 4 mm), mild pain (5- 44), moderate pain (45-74 mm), and severe pain (75- 100 mm).
  Patients were also asked to take analgesic (ibuprofen 400 mg/6-8h) according to the intensity of pain experienced by them and note down the details of analgesic intake on the proforma regarding the number of doses required and timing of the dose.

IPD SHARING:
Plan to Share IPD: No